CLINICAL TRIAL: NCT00843128
Title: Phase II Study of the Effectiveness of Locomotor Therapy Using Robot-Driven Gait Orthosis System in Acute Stroke Patients: A Randomized Controlled Trial.
Brief Title: The Effectiveness of Locomotor Therapy Using Robot-Driven Gait Orthosis System in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Zeev Meiner, Hadassah Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0558-08-HMO-CTIL
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2009-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: RAGT (Experimental): Following randomization, 20 patients will be treated with RAGT, 12 sessions over three weeks
  Interventions: Device: robot-assisted gait training (RAGT)
- 2: Control (Active Comparator): The control group will be treated by CWT, 12 sessions in three weeks.
  Interventions: Device: conventional walking training (CWT)

INTERVENTIONS:
Device: robot-assisted gait training (RAGT) — 20 patients will be treated with RAGT, 12 sessions over three weeks.
  Arms: 1: RAGT
Device: conventional walking training (CWT) — The control group will be treated by CWT, 12 sessions in three weeks.
  Arms: 2: Control

SUMMARY:
Objective: To evaluate the efficacy of robot-assisted gait training (RAGT) in MS patients with severe walking disabilities (Expanded Disability Status Scale [EDSS] 5.5-7) as compared to regular physiotherapy.

Methods: Prospective, randomized, controlled clinical trial comparing RAGT with conventional walking training (CWT) in a group of stable MS patients (n=40) during an outpatient rehabilitation program. Inclusion criteria are chronic or secondary progressive MS patients with EDSS between 5.5-7, stable treatment 3 months before study entry, without generalized diseases. All patients will sign an informed consent. Following randomization, 20 patients will be treated with RAGT, 12 sessions over three weeks. The control group will be treated by CWT, 12 sessions in three weeks. The primary outcome measures will be the Functional Ambulatory Capacity (FAC) scale and the 6-minutes walking distance. The secondary outcome measures will be the Time up & Go (TUG) test, 10 Meter Walking test, Berg balance test, EDSS score, FIM score and RAND questioner for quality of life. All tests will be performed by an external blinded assessor at baseline, after three weeks, and at follow-up after 3 months and six months.

Importance: We anticipated that Robot-assisted gait training will be found as feasible and may be an effective therapeutic option in MS patients with severe walking disabilities.

ELIGIBILITY:
Inclusion Criteria:

1. chronic or secondary progressive MS patients with EDSS between 5.5-7,
2. stable treatment 3 months before study entry.

Exclusion Criteria:

1. Other generalized diseases.
2. Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Functional Ambulatory Capacity (FAC) scale and the 6-minutes walking distance | At baseline, after three weeks, and at follow-up after 3 months and six months.

SECONDARY OUTCOMES:
Time up & Go (TUG) test, 10 Meter Walking test, Berg balance test, EDSS score, FIM score and SF36 questioner for quality of life. | At baseline, after three weeks, and at follow-up after 3 months and six months.

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Meiner, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel